CLINICAL TRIAL: NCT05332106
Title: Bioavailability of a Formulation of Estradiol Valerate and Dienogest 2 mg/2 mg Coated Tablets With Regards to the Marketed Reference Product
Brief Title: Bioavailability of Estradiol Valerate and Dienogest 2 mg/2 mg With Regards to Reference Product
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratorios Andromaco S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HP8833-01
Record Dates: First submitted 2022-04-05; First posted 2022-04-18 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Bioequivalence
MeSH Terms: interventions — Estradiol; dienogest; Drug Evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Estradiol Valerate and Dienogest Test Product. (Experimental): Participants will receive one tablet of the test formulation containing Estradiol Valerate and Dienogest 2 mg/ 2 mg.The tablet will be taken with water and in a fasting condition.
  Interventions: Drug: Estradiol Valerate and Dienogest 2 mg/ 2 mg Test Drug tablet
- Estradiol Valerate and Dienogest Referent Product (Active Comparator): Participants will receive one tablet of the marketed reference containing Estradiol Valerate and Dienogest 2 mg/ 2 mg. The tablet will be taken with water and in a fasting condition.
  Interventions: Drug: Estradiol Valerate and Dienogest 2 mg/ 2 mg Reference Product tablet

INTERVENTIONS:
Drug: Estradiol Valerate and Dienogest 2 mg/ 2 mg Test Drug tablet — Investigational Medicinal Product
  Arms: Estradiol Valerate and Dienogest Test Product.
Drug: Estradiol Valerate and Dienogest 2 mg/ 2 mg Reference Product tablet — Climodien (Bayer plc.)
  Arms: Estradiol Valerate and Dienogest Referent Product

SUMMARY:
This study will investigate the bioavailability in fasting healthy, adult, human post-menopausal female subjects of 1 tablet formulation containing Estradiol Valerate and Dienogest 2 mg/ 2mg.

The study will be performed at a single site with 10 subjects. Participants will take 1 tablet of the test product and reference product in 2 periods and 2 sequences (either test after reference or reference after test). There will be a washout of at least 7 days between each study period.

DETAILED DESCRIPTION:
The primary objective of the study is to investigate the relative bioavailability of Estradiol Valerate and Dienogest 2mg/ 2mg of 1 tablet formulations with Estradiol Valerate and Dienogest 2mg/ 2mg and to demonstrate bioequivalence of both formulations in terms of rate and extent of absorption:

* Test Product: Product manufactured by Laboratorios Andromaco S.A.
* Reference Product: Climodien [Trademark], product Bayer plc. The 90% confidence intervals for the intra-subject coefficient of variation (Test versus Reference Product) for the main pharmacokinetic parameters area under the plasma concentration-time curve from time zero to time t (AUC0 0-t) and from time zero to infinite (AUC0 0-∞), and maximum plasma concentration (Cmax) for total Estradiol and Dienogest will be determined. Participants will be confined in the study site for approximately 42 hours during the entire study (for 10 hours pre-dosing and for 32 hours post dosing in both periods) during which pharmacokinetic (PK) blood samples will be obtained. 26 blood samples will be taken up to 72 hours after the administration in each period. The washout period between the two study periods will be at least 7 days. The samples from each participant will be analyzed with validated LC-MS/MS method for estimation of Estradiol and Dienogest in plasma. The safety objective is to evaluate the tolerability of both formulations in subjects by collecting adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy post-menopausal female literate volunteers of 40 to 65 years (both years inclusive) with BMI of 18.50 - 29.99 Kg/m2 and weight > 50 Kg.
2. Healthy volunteers as evaluated by medical history, vitals and general clinical examination.
3. Normal or clinically insignificant biochemical, hematological, urine and serology parameters.
4. Normal or clinically insignificant ECG.
5. Negative urine test for drugs of abuse and negative pregnancy test.
6. Volunteers who are willing to use acceptable methods of contraception (barrier method/IUD/surgical) or abstinence, for the entire duration of the study and do not plan to be pregnant for at least 1 month after the last drug administration.
7. Volunteers who can give written informed consent and communicate effectively.

Exclusion Criteria:

1. History of any major surgical procedure in the past 03 months.
2. History of any clinically significant cardiac, gastrointestinal, respiratory, hepatic, renal, endocrine, neurological, metabolic, psychiatric and hematological disorders.
3. History of chronic alcoholism/ chronic smoking/ drug of abuse.
4. Volunteers with known hypersensitivity to Dienogest/Estradiol Valerate or any of the excipients.
5. History of consumption of tobacco containing products within 48 hours prior to proposed time of dosing.
6. Volunteers who are positive for hepatitis B surface antigen, anti-hepatitis C antibody, treponemal antibodies and human immunodeficiency virus (HIV 1&2) antibodies.
7. Present or past history of intake of drugs or any prescription drug or over the counter (OTC) drugs within 14 days which potentially modify kinetics / dynamics of Dienogest/Estradiol Valerate or any other medication judged to be clinically significant by the investigator.
8. History of consumption of grapefruit and/or its products within 10 days prior to the start of study.
9. Volunteers who had participated in any other clinical study or who had bled during the last 03 months before check-in.
10. History of consumption of one or more of the below, 48 hours prior to dosing: Xanthine containing food or drinks such as cola, chocolate, coffee or tea, citrus fruits or items (lime, lemon and orange), alcohol and any other food/beverage known to have interactions as deemed by the investigator.
11. Volunteers who are dysphagic.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-03-12 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2022-03-22 (Actual)

PRIMARY OUTCOMES:
Total Estradiol Valerate: area under the plasma concentration-time curve from 0 to time t (AUC0-72) | From tablet intake and up to 72 hours after tablet intake
  26 samples up to 72 hours will be taken after the administration in each period
Total Estradiol Valerate: Maximum plasma concentration (Cmax) | From tablet intake and up to 72 hours after tablet intake
  26 samples up to 72 hours will be taken after the administration in each period
Total Estradiol Valerate: Time to achieve maximum plasma concentration (tmax) | From tablet intake and up to 72 hours after tablet intake
  26 samples up to 72 hours will be taken after the administration in each period
Total Dienogest: area under the plasma concentration-time curve from 0 to time t (AUC0-72) | From tablet intake and up to 72 hours after tablet intake
  26 samples up to 72 hours will be taken after the administration in each period
Total Dienogest: Maximum plasma concentration (Cmax) | From tablet intake and up to 72 hours after tablet intake
  26 samples up to 72 hours will be taken after the administration in each period
Total Dienogest: Time to achieve maximum plasma concentration (tmax) | From tablet intake and up to 72 hours after tablet intake
  26 samples up to 72 hours will be taken after the administration in each period

CONTACTS AND LOCATIONS:
Overall Officials: R. Amirtha, MD, Principal Investigator — Azidus Laboratories Ltd.
Locations (1):
- Azidus Laboratories Ltd., Chennai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No